CLINICAL TRIAL: NCT01567085
Title: An Open-Label, Single-Arm, Multicenter Trial to Determine Safety and Efficacy of Eculizumab in the Prevention of Antibody Mediated Rejection (AMR) in Sensitized Recipients of a Kidney Transplant From a Deceased Donor.
Brief Title: Safety & Efficacy Of Eculizumab In The Prevention Of AMR In Sensitized Recipients Of A Kidney Transplant From A Deceased Donor
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Alexion Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: C10-002; 2010-019631-35 (EudraCT Number)
Record Dates: First submitted 2012-03-27; First posted 2012-03-30 (Estimated); Results first posted 2019-05-03 (Actual); Last update posted 2019-05-03 (Actual); Status verified 2019-01

CONDITIONS: Stage V Chronic Kidney Disease
MeSH Terms: interventions — eculizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Eculizumab (Experimental): Eculizumab 1200 milligrams (mg) was administered intravenously (IV) over 25 to 45 minutes 1 hour prior to kidney allograft reperfusion.
  Eculizumab 900 mg was administered IV over 25 to 45 minutes on post-transplantation Days 1 and 7, and on post-transplantation Days 14, 21, and 28, plus or minus 2 days.
  Eculizumab 1200 mg was administered IV over 25 to 45 minutes on post-transplantation Days 35, 49, and 63, plus or minus 2 days.
  Interventions: Drug: Eculizumab

INTERVENTIONS:
Drug: Eculizumab
  Other Names: Soliris

SUMMARY:
Primary Objective:

To evaluate the safety and potential efficacy of eculizumab to prevent AMR in sensitized recipients of deceased donor kidney transplants.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female participants ≥18 years old.
2. Participants with Stage V chronic kidney disease who received a kidney transplant from a deceased donor to whom they were sensitized.
3. History of prior exposure to HLA (human leukocyte antigen):

   * Prior solid organ or tissue allograft
   * Pregnancy
   * Blood transfusion
   * Prior exposure to specific donor's HLA

Exclusion Criteria:

1. Has received treatment with eculizumab at any time prior to enrolling in this study.
2. Blood type (A, B, and O blood glycoproteins-blood type) incompatible with deceased donor.
3. History of severe cardiac disease.
4. Prior splenectomy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2012-08-29 (Actual); Primary Completion 2015-06-11 (Actual); Study Completion 2017-05-24 (Actual)

CONTACTS AND LOCATIONS:
Locations (14):
- Australia (3):
  - Adelaide
  - Camperdown
  - Parkville
- France (4):
  - Bordeaux
  - Paris
  - Toulouse
  - Tours
- Italy (2):
  - Brescia
  - Padua
- Barcelona, Spain
- Sweden (2):
  - Gothenburg
  - Uppsala
- United Kingdom (2):
  - Cambridge
  - London

RESULTS

PARTICIPANT FLOW:
Groups:
- Eculizumab: All eculizumab was administered intravenously (IV) over 25 to 45 minutes. Eculizumab 1200 milligrams (mg) was administered approximately 1 hour prior to kidney allograft reperfusion.
  Eculizumab 900 mg was administered IV over 25 to 45 minutes on post-transplantation Days 1 and 7, and on post-transplantation Days 14, 21, and 28, plus or minus 2 days.
  Eculizumab 1200 mg was administered IV over 25 to 45 minutes on post-transplantation Days 35, 49, and 63, plus or minus 2 days.
Period: Overall Study
Arm/Group | Eculizumab
Started | 80
Received at Least 1 Dose of Study Drug | 80
Completed | 60
Not Completed | 20
Not completed — Death | 6
Not completed — Adverse Event | 6
Not completed — Lost to Follow-up | 3
Not completed — Graft loss | 2
Not completed — Renal transplantectomy | 1
Not completed — Returned to chronic dialysis | 1
Not completed — Terminal chronic kidney dysfunction | 1

BASELINE CHARACTERISTICS:
Population: Safety Population: enrolled participants who received at least 1 dose of eculizumab.
Groups:
- Eculizumab: All eculizumab was administered IV over 25 to 45 minutes. Eculizumab 1200 mg was administered approximately 1 hour prior to kidney allograft reperfusion.
  Eculizumab 900 mg was administered IV over 25 to 45 minutes on post-transplantation Days 1 and 7, and on post-transplantation Days 14, 21, and 28, plus or minus 2 days.
  Eculizumab 1200 mg was administered IV over 25 to 45 minutes on post-transplantation Days 35, 49, and 63, plus or minus 2 days.
Arm/Group | Eculizumab
Number analyzed (Participants) | 80
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.7 (11.26)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 48
  Male | 32
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 5
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 7
  White | 59
  Unknown or Not Reported | 9

OUTCOME MEASURES:

1. Primary Outcome: Post-transplantation Treatment Failure In The First 9 Weeks Post Transplantation
Description: Results are reported for post-transplantation treatment failure and composite endpoints, defined as the occurrence of biopsy-proven acute antibody-mediated rejection (AMR), graft loss, death, or loss to follow-up (including discontinuation) in the first 9 weeks post transplantation. The diagnosis of acute AMR (occurring within the first 9 weeks post transplantation) was based on kidney allograft dysfunction and a biopsy performed due to suspected rejection, proteinuria, increased serum creatinine, or acute tubular necrosis. Treatment failure was the occurrence of at least 1 of the composite endpoint components by Week 9 post transplantation. A participant experiencing multiple events was only counted once for the composite endpoint.
Time Frame: Baseline, Week 9
Population: Full Analysis Population: participants who were enrolled, received a deceased donor kidney transplant, and received at least 1 dose of eculizumab.
Measure: Count of Participants; unit: Participants
Arm/Group | Eculizumab
Number analyzed (Participants) | 80
Participants
  Treatment Failure - Yes | 7
  Treatment Failure - No | 73
  Biopsy-proven Acute AMR | 3
  Graft Loss | 4
  Death | 1
  Lost to Follow-up (Including Discontinuation) | 1
Statistical Analysis 1: Comparison: Eculizumab; Analysis of post-transplantation treatment failure rate; Test type: Other — Exact binomial test; p < 0.001, Exact binomial test — The p-value was calculated from an exact binomial test, where the null hypothesis was that the true failure rate = 40%; Exact 95% confidence interval (3.6, 17.2)

2. Other Pre Specified Outcome: Cumulative Incidence Function (CIF) Of Other Adverse Events (AEs) Of Interest At Month 12
Description: Specific analyses of other AEs of interest that occurred at Month 12 included cumulative incidence of clinically significant infection (CSI); post-transplant lymphoproliferative disease (PTLD); malignancies; biopsy-proven acute cellular rejection (ACR) of any grade meeting Banff 2007 criteria; allograft loss for reasons other than AMR. CSIs were defined as infections (confirmed by culture, biopsy, genomic, or serologic findings) that required hospitalization or anti-infective treatment, or otherwise deemed significant by the Investigator. CSI subcategories of interest included cytomegalovirus (CMV) disease; BK virus disease; encapsulated bacterial infection; fungal infections; aspergillus infections. Results are reported as CIF, where a larger CIF indicates a higher incidence of an AE, and were calculated using Statistical Analysis System software and macro CIF. A summary of serious and all other non-serious AEs regardless of causality is located in the Reported Adverse Events module.
Time Frame: Baseline, Month 12
Population: Safety Population: enrolled participants who received at least 1 dose of eculizumab.
Measure: Number (95% Confidence Interval); unit: Proportion of Adverse Events
Arm/Group | Eculizumab
Number analyzed (Participants) | 80
Proportion of Adverse Events
  Confirmed CSI | 0.7989 [0.69 to 0.87]
  CMV Infection | 0.2994 [0.20 to 0.40]
  BK Virus Infection | 0.1536 [0.08 to 0.24]
  Encapsulated Bacterial Infection | 0.1642 [0.09 to 0.25]
  Fungal Infection | 0.1287 [0.07 to 0.21]
  Aspergillus Infection | 0 [0 to 0]
  PTLD | 0.0264 [0.00 to 0.08]
  Malignancies | 0.0264 [0.00 to 0.08]
  Biopsy-proven ACR | 0.0375 [0.01 to 0.10]
  Allograft Loss For Reasons Other Than AMR | 0.1132 [0.06 to 0.19]

3. Other Pre Specified Outcome: Participants That Developed Severe ACR (Other AE Of Interest) At Month 12
Description: This outcome measure focuses on the other AE of interest, severe ACR, which occurred at Month 12. It pertains specifically to the number of participants who developed severe ACR that did not respond to thymoglobulin or other lymphocyte-depleting agents. A summary of serious and all other non-serious AEs, regardless of causality, is located in the Reported Adverse Events module.
Time Frame: Baseline, Month 12
Population: Safety Population: participants who received at least 1 dose of eculizumab.
Measure: Count of Participants; unit: Participants
Arm/Group | Eculizumab
Number analyzed (Participants) | 80
Participants | 3

ADVERSE EVENTS:
Time Frame: Adverse event data were collected beginning on the day of transplantation, Day 0, through 12 months post transplantation.
Arm/Group | Eculizumab
All-Cause Mortality (participants affected / at risk) | 6/80
Serious Adverse Events (participants affected / at risk) | 70/80
Other Adverse Events (participants affected / at risk) | 80/80
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Eculizumab (N=80)
Anaemia (Blood and lymphatic system disorders) | 4
Febrile neutropenia (Blood and lymphatic system disorders) | 2
Leukopenia (Blood and lymphatic system disorders) | 3
Neutropenia (Blood and lymphatic system disorders) | 1
Pancytopenia (Blood and lymphatic system disorders) | 4
Thrombotic microangiopathy (Blood and lymphatic system disorders) | 1
Angina pectoris (Cardiac disorders) | 1
Atrial fibrillation (Cardiac disorders) | 1
Atrioventricular block complete (Cardiac disorders) | 1
Myocardial ischaemia (Cardiac disorders) | 1
Supraventricular tachycardia (Cardiac disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 2
Ascites (Gastrointestinal disorders) | 1
Colitis (Gastrointestinal disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 4
Gingivitis ulcerative (Gastrointestinal disorders) | 1
Impaired gastric emptying (Gastrointestinal disorders) | 1
Inguinal hernia (Gastrointestinal disorders) | 1
Intestinal obstruction (Gastrointestinal disorders) | 2
Intra-abdominal fluid collection (Gastrointestinal disorders) | 1
Palatal disorder (Gastrointestinal disorders) | 1
Pneumoperitoneum (Gastrointestinal disorders) | 1
Rectal haemorrhage (Gastrointestinal disorders) | 1
Small intestinal obstruction (Gastrointestinal disorders) | 1
Small intestinal perforation (Gastrointestinal disorders) | 1
Umbilical hernia (Gastrointestinal disorders) | 1
Catheter site pain (General disorders) | 1
Chest pain (General disorders) | 1
Multiple organ dysfunction syndrome (General disorders) | 1
Non-cardiac chest pain (General disorders) | 1
Pyrexia (General disorders) | 2
Ulcer haemorrhage (General disorders) | 1
Cholangitis (Hepatobiliary disorders) | 1
Cholecystitis (Hepatobiliary disorders) | 1
Cholecystitis acute (Hepatobiliary disorders) | 1
Cholelithiasis (Hepatobiliary disorders) | 1
Drug-induced liver injury (Hepatobiliary disorders) | 1
Jaundice cholestatic (Hepatobiliary disorders) | 1
Drug hypersensitivity (Immune system disorders) | 1
Kidney transplant rejection (Immune system disorders) | 25
BK virus infection (Infections and infestations) | 1
Bacteraemia (Infections and infestations) | 1
Bacterial pyelonephritis (Infections and infestations) | 5
Bronchitis (Infections and infestations) | 1
Bronchitis viral (Infections and infestations) | 1
Campylobacter infection (Infections and infestations) | 1
Candiduria (Infections and infestations) | 1
Catheter site infection (Infections and infestations) | 1
Clostridium difficile colitis (Infections and infestations) | 1
Cytomegalovirus colitis (Infections and infestations) | 1
Cytomegalovirus infection (Infections and infestations) | 5
Device related sepsis (Infections and infestations) | 1
Diarrhoea infectious (Infections and infestations) | 1
Encephalitis (Infections and infestations) | 1
Enterococcal sepsis (Infections and infestations) | 1
Escherichia pyelonephritis (Infections and infestations) | 4
Escherichia sepsis (Infections and infestations) | 2
Escherichia urinary tract infection (Infections and infestations) | 4
Gastroenteritis (Infections and infestations) | 4
Gastroenteritis norovirus (Infections and infestations) | 4
Gastroenteritis viral (Infections and infestations) | 1
Gingival abscess (Infections and infestations) | 1
Haematoma infection (Infections and infestations) | 1
Hepatic cyst infection (Infections and infestations) | 1
Hepatitis C (Infections and infestations) | 1
Incision site infection (Infections and infestations) | 1
Infected cyst (Infections and infestations) | 1
Infected fistula (Infections and infestations) | 1
Klebsiella infection (Infections and infestations) | 1
Klebsiella sepsis (Infections and infestations) | 2
Lung abscess (Infections and infestations) | 1
Periodontitis (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 5
Pneumonia cryptococcal (Infections and infestations) | 1
Polyomavirus-associated nephropathy (Infections and infestations) | 3
Pyelonephritis (Infections and infestations) | 7
Pyelonephritis acute (Infections and infestations) | 2
Sepsis (Infections and infestations) | 2
Septic shock (Infections and infestations) | 1
Systemic mycosis (Infections and infestations) | 1
Tooth infection (Infections and infestations) | 1
Upper respiratory tract infection (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 3
Urinary tract infection bacterial (Infections and infestations) | 2
Urosepsis (Infections and infestations) | 3
Viral infection (Infections and infestations) | 1
Accidental overdose (Injury, poisoning and procedural complications) | 2
Arteriovenous fistula thrombosis (Injury, poisoning and procedural complications) | 3
Complications of transplanted kidney (Injury, poisoning and procedural complications) | 4
Delayed graft function (Injury, poisoning and procedural complications) | 10
Fall (Injury, poisoning and procedural complications) | 1
Incisional hernia (Injury, poisoning and procedural complications) | 1
Post procedural haematoma (Injury, poisoning and procedural complications) | 3
Post procedural haematuria (Injury, poisoning and procedural complications) | 2
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 4
Traumatic haematoma (Injury, poisoning and procedural complications) | 1
Urinary anastomotic leak (Injury, poisoning and procedural complications) | 1
Wound (Injury, poisoning and procedural complications) | 1
Antibody test positive (Investigations) | 2
Blood creatinine increased (Investigations) | 6
White blood cell count increased (Investigations) | 1
Calciphylaxis (Metabolism and nutrition disorders) | 1
Dehydration (Metabolism and nutrition disorders) | 1
Diabetes mellitus (Metabolism and nutrition disorders) | 4
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 2
Hypercalcaemia (Metabolism and nutrition disorders) | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 3
Hypoglycaemia (Metabolism and nutrition disorders) | 1
Hyponatraemia (Metabolism and nutrition disorders) | 2
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1
Ductal adenocarcinoma of pancreas (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Medullary thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Metastatic squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Neuroendocrine tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Refractory anaemia with an excess of blasts (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Disturbance in attention (Nervous system disorders) | 1
Headache (Nervous system disorders) | 1
Loss of consciousness (Nervous system disorders) | 1
Migraine (Nervous system disorders) | 1
Seizure (Nervous system disorders) | 1
Toxic encephalopathy (Nervous system disorders) | 1
Pre-eclampsia (Pregnancy, puerperium and perinatal conditions) | 1/48
Premature delivery (Pregnancy, puerperium and perinatal conditions) | 1/48
Acute kidney injury (Renal and urinary disorders) | 12
Anuria (Renal and urinary disorders) | 1
Haematuria (Renal and urinary disorders) | 5
Hydronephrosis (Renal and urinary disorders) | 3
Proteinuria (Renal and urinary disorders) | 1
Renal artery thrombosis (Renal and urinary disorders) | 2
Renal cyst (Renal and urinary disorders) | 1
Renal cyst haemorrhage (Renal and urinary disorders) | 1
Renal failure (Renal and urinary disorders) | 1
Renal haematoma (Renal and urinary disorders) | 1
Renal impairment (Renal and urinary disorders) | 3
Renal tubular necrosis (Renal and urinary disorders) | 1
Renal vascular thrombosis (Renal and urinary disorders) | 1
Renal vein thrombosis (Renal and urinary disorders) | 1
Urinoma (Renal and urinary disorders) | 1
Vaginal dysplasia (Reproductive system and breast disorders) | 1/48
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 5
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1
Skin ulcer (Skin and subcutaneous tissue disorders) | 1
Plastic surgery (Surgical and medical procedures) | 1
Arterial disorder (Vascular disorders) | 1
Arteriovenous fistula (Vascular disorders) | 1
Deep vein thrombosis (Vascular disorders) | 1
Hypertension (Vascular disorders) | 1
Hypotension (Vascular disorders) | 2
Lymphocele (Vascular disorders) | 2
Peripheral artery thrombosis (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Eculizumab (N=80)
Anaemia (Blood and lymphatic system disorders) | 51
Leukopenia (Blood and lymphatic system disorders) | 30
Lymphopenia (Blood and lymphatic system disorders) | 11
Neutropenia (Blood and lymphatic system disorders) | 18
Pancytopenia (Blood and lymphatic system disorders) | 7
Thrombocytopenia (Blood and lymphatic system disorders) | 12
Palpitations (Cardiac disorders) | 5
Tachycardia (Cardiac disorders) | 6
Abdominal pain (Gastrointestinal disorders) | 14
Abdominal pain upper (Gastrointestinal disorders) | 9
Constipation (Gastrointestinal disorders) | 15
Diarrhoea (Gastrointestinal disorders) | 37
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 12
Mouth ulceration (Gastrointestinal disorders) | 7
Nausea (Gastrointestinal disorders) | 25
Vomiting (Gastrointestinal disorders) | 18
Asthenia (General disorders) | 13
Chest pain (General disorders) | 7
Influenza like illness (General disorders) | 9
Oedema (General disorders) | 5
Oedema peripheral (General disorders) | 31
Pyrexia (General disorders) | 20
Cholestasis (Hepatobiliary disorders) | 6
Hypogammaglobulinaemia (Immune system disorders) | 5
Kidney transplant rejection (Immune system disorders) | 22
BK virus infection (Infections and infestations) | 10
Bacterial pyelonephritis (Infections and infestations) | 5
Bronchitis (Infections and infestations) | 9
Conjunctivitis (Infections and infestations) | 5
Escherichia infection (Infections and infestations) | 8
Escherichia urinary tract infection (Infections and infestations) | 8
Gastroenteritis (Infections and infestations) | 7
Gastroenteritis norovirus (Infections and infestations) | 6
Nasopharyngitis (Infections and infestations) | 11
Oral candidiasis (Infections and infestations) | 6
Pneumonia (Infections and infestations) | 4
Polyomavirus-associated nephropathy (Infections and infestations) | 4
Pyelonephritis (Infections and infestations) | 10
Upper respiratory tract infection (Infections and infestations) | 10
Urinary tract infection (Infections and infestations) | 32
Accidental overdose (Injury, poisoning and procedural complications) | 5
Arteriovenous fistula thrombosis (Injury, poisoning and procedural complications) | 5
Complications of transplanted kidney (Injury, poisoning and procedural complications) | 5
Delayed graft function (Injury, poisoning and procedural complications) | 12
Post procedural haematoma (Injury, poisoning and procedural complications) | 6
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 5
Procedural pain (Injury, poisoning and procedural complications) | 11
Blood creatinine increased (Investigations) | 15
Cardiac murmur (Investigations) | 5
Liver function test abnormal (Investigations) | 8
Weight decreased (Investigations) | 7
Weight increased (Investigations) | 5
Acidosis (Metabolism and nutrition disorders) | 21
Decreased appetite (Metabolism and nutrition disorders) | 6
Dehydration (Metabolism and nutrition disorders) | 5
Diabetes mellitus (Metabolism and nutrition disorders) | 11
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 4
Fluid overload (Metabolism and nutrition disorders) | 9
Hypercalcaemia (Metabolism and nutrition disorders) | 8
Hyperglycaemia (Metabolism and nutrition disorders) | 14
Hyperkalaemia (Metabolism and nutrition disorders) | 23
Hyperphosphataemia (Metabolism and nutrition disorders) | 10
Hypocalcaemia (Metabolism and nutrition disorders) | 14
Hypoglycaemia (Metabolism and nutrition disorders) | 8
Hypokalaemia (Metabolism and nutrition disorders) | 18
Hypomagnesaemia (Metabolism and nutrition disorders) | 16
Hyponatraemia (Metabolism and nutrition disorders) | 9
Hypophosphataemia (Metabolism and nutrition disorders) | 11
Vitamin D deficiency (Metabolism and nutrition disorders) | 8
Back pain (Musculoskeletal and connective tissue disorders) | 12
Muscle spasms (Musculoskeletal and connective tissue disorders) | 5
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 19
Headache (Nervous system disorders) | 22
Tremor (Nervous system disorders) | 7
Anxiety (Psychiatric disorders) | 9
Insomnia (Psychiatric disorders) | 9
Acute kidney injury (Renal and urinary disorders) | 10
Dysuria (Renal and urinary disorders) | 8
Haematuria (Renal and urinary disorders) | 11
Proteinuria (Renal and urinary disorders) | 16
Renal impairment (Renal and urinary disorders) | 9
Renal tubular necrosis (Renal and urinary disorders) | 13
Urinary incontinence (Renal and urinary disorders) | 8
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 6
Cough (Respiratory, thoracic and mediastinal disorders) | 18
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 19
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 5
Rales (Respiratory, thoracic and mediastinal disorders) | 6
Pruritus (Skin and subcutaneous tissue disorders) | 8
Deep vein thrombosis (Vascular disorders) | 4
Haematoma (Vascular disorders) | 6
Hypertension (Vascular disorders) | 31
Hypotension (Vascular disorders) | 13
Lymphocele (Vascular disorders) | 5
Orthostatic hypotension (Vascular disorders) | 6
Cytomegalovirus infection (Infections and infestations) | 21
Hypercholesterolaemia (Metabolism and nutrition disorders) | 6
Alopecia (Skin and subcutaneous tissue disorders) | 5
Clostridium difficile infection (Infections and infestations) | 4
Ear infection (Infections and infestations) | 4
Enterococcal infection (Infections and infestations) | 4
Escherichia pyelonephritis (Infections and infestations) | 4
Herpex simplex (Infections and infestations) | 4
Sinusitis (Infections and infestations) | 4
Urinary tract infection bacterial (Infections and infestations) | 4
Cell death (Metabolism and nutrition disorders) | 4
Hyperlipidaemia (Metabolism and nutrition disorders) | 4
Dyspepsia (Gastrointestinal disorders) | 4
Gastritis (Gastrointestinal disorders) | 4
Haemorrhoids (Gastrointestinal disorders) | 4
Oliguria (Renal and urinary disorders) | 4
Polyuria (Renal and urinary disorders) | 4
Renal artery stenosis (Renal and urinary disorders) | 4
Pain (General disorders) | 4
Incisional hernia (Injury, poisoning and procedural complications) | 4
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 4
Productive cough (Respiratory, thoracic and mediastinal disorders) | 4
Dizziness (Nervous system disorders) | 4
Depression (Psychiatric disorders) | 4
Atrial fibrillation (Cardiac disorders) | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2013-10-08): https://cdn.clinicaltrials.gov/large-docs/85/NCT01567085/Prot_000.pdf
  • Statistical Analysis Plan (2013-11-12): https://cdn.clinicaltrials.gov/large-docs/85/NCT01567085/SAP_001.pdf